CLINICAL TRIAL: NCT05459350
Title: Prediction of Safe Discharge From ICU
Acronym: SAFEDI
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SAFEDI
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Safe Discharge Positive: Safe Discharge Positive
  Interventions: Diagnostic Test: Safe Discharge Classification
- Safe Discharge Negative: Safe Discharge Negative
  Interventions: Diagnostic Test: Safe Discharge Classification

INTERVENTIONS:
Diagnostic Test: Safe Discharge Classification — Safe Discharge Classification

SUMMARY:
Patients who have an increased need for monitoring or therapy during their stay in hospital are typically admitted to an intensive care unit. This is characterized by a large number of diagnostic and therapeutic options. If this additional effort is no longer necessary, then typically in most hospitals patients are transferred to wards with a lower presence of nurses and physicians and reduced provision of extensive monitoring and therapeutic procedures such as organ replacement procedures.

However, deintensification of medical and nursing care requires that previously monitored and partially supported bodily functions are restored to the point where further monitoring is no longer necessary. For this reason, transfer from an intensive care unit to the normal inpatient area is only possible if the patient in question has neither an increased need for monitoring nor an increased need for therapy. If this is not the case, then there is a risk of life-threatening conditions in the normal ward, which can sometimes occur very quickly. However, the need for further monitoring, or for continued intensive medical therapy, cannot be easily assessed. There is no laboratory value or clinical examination method that can be used to estimate beyond doubt whether a patient's condition could worsen if he or she is transferred to the normal ward. For this reason, the decision to transfer is made on the basis of the individual assessment by the attending physician. Although this is based on the synopsis of a wide variety of examinations and laboratory findings, it is therefore subject to large interindividual variations. Thus, the personal experience of the evaluating physician has a considerable influence on the decision for or against a transfer to the normal inpatient area.

In this respect, the decision to deintensify therapy, i.e. to transfer patients from intensive care units to the normal care area, is challenging:

The assessing physician has to make a prediction from the combination of the available findings under time pressure whether a transfer to the normal inpatient area is possible without endangering the patient. In this situation, it would be desirable to have an automated warning system that could describe the success of the transfer with sufficient accuracy in the presence of specific laboratory constellations. In the best case, such an approach would prevent dangerous transfers, but at the same time reduce unnecessary lengths of stay in the ICU. Machine learning methods seem particularly suited to support such a decision.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients that were treated in intensive care units at the Kepler University Hospital in Linz, Austria in the period 2010-01-01 to 2019-10-31.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As described in the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 24010 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
AUROC for Classification of Safe Discharge | 2010-01-01 to 2019-10-31
  AUROC for Classification of Safe Discharge

SECONDARY OUTCOMES:
Confusion Matrix Value | 2010-01-01 to 2019-10-31
  Confusion Matrix Results: true positives, true negatives, false positive, false negatives and values calculated from these results.
Descriptive Statistics | 2010-01-01 to 2019-10-31
  Descriptive Statistics (age in years, height in cm, weight in kg, gender as male/female, date of death, standard laboratory measurements (e. g. blood gas analysis, full blood count, liver function tests, kidney function tests), ICD 10-codes associated with the patient's admission, Glasgow Coma Scale)
  This outcome measure will compare the individual feature (e. g. height in cm) in one group vs. the other. Significant difference will be described by p-value.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tschoellitsch, MD, Principal Investigator — Kepler University Hospital and Johannes Kepler University, Linz, Austria
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No